CLINICAL TRIAL: NCT03805035
Title: Anti-histamines Promote Electroacupuncture Analgesia: Basic and Clinical Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CMUH107-REC3-019
Record Dates: First submitted 2019-01-08; First posted 2019-01-15 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Pain
Keywords: Electroacupuncture (EA); Antihistamine; Pain
MeSH Terms: conditions — Pain | interventions — Electroacupuncture; Histamine Antagonists; Chlorpheniramine; dexchlorpheniramine; Tablets; Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- sham EA group (Sham Comparator): Minimal needling at ST36 and GB34 (n=10)
  Interventions: Device: acupuncture
- true EA group (Experimental): EA at ST36 and GB34 (n=10)
  Interventions: Device: electroacupuncture
- EA+antihistamine(low dose) group (Active Comparator): EA at ST36 and GB34 plus low-dose chlorpheniramine( Dexchlorpheniramine maleate 2mg/tab, 1 tab; n=10)
  Interventions: Device: electroacupuncture; Drug: antihistamine(low dose) chlorpheniramine (Dexchlorpheniramine maleate)
- EA+antihistamine(high dose) group (Active Comparator): EA at ST36 and GB34 plus high-dose chlorpheniramine (Dexchlorpheniramine maleate 2mg/tab, 2 tabs; n=10)
  Interventions: Device: electroacupuncture; Drug: antihistamine(high dose) chlorpheniramine (Dexchlorpheniramine maleate)

INTERVENTIONS:
Device: electroacupuncture — Group 2 (n=10) EA at ST36 and GB34;intensity (2 mA), pulse width (1 ms), frequency (2 Hz)
  Arms: EA+antihistamine(high dose) group; EA+antihistamine(low dose) group; true EA group
Drug: antihistamine(low dose) chlorpheniramine (Dexchlorpheniramine maleate) — Group 3 (n=10) EA at ST36 and GB34 plus chlorpheniramine (Dexchlorpheniramine maleate 2mg/tab, 1 tab);intensity (2 mA), pulse width (1 ms), frequency (2 Hz)
  Other Names: chlorpheniramine (Dexchlorpheniramine maleate 2mg/tab, 1 tab)
  Arms: EA+antihistamine(low dose) group
Drug: antihistamine(high dose) chlorpheniramine (Dexchlorpheniramine maleate) — Group 4 (n=10) EA at ST36 and GB34 plus chlorpheniramine (Dexchlorpheniramine maleate2mg/tab, 2 tabs);intensity (2 mA), pulse width (1 ms), frequency (2 Hz)
  Other Names: chlorpheniramine (Dexchlorpheniramine maleate2mg/tab, 2 tabs)
  Arms: EA+antihistamine(high dose) group
Device: acupuncture — Minimal needling at ST36 and GB34
  Other Names: shallow needling
  Arms: sham EA group

SUMMARY:
Acupuncture has been used in traditional Chinese medicine for around 3,000 years and is increasingly practiced worldwide. The effects of acupuncture in chronic pain have been investigated in many clinical trials. Histamine H1 receptor antagonists are commonly used for treating allergy. Recently, investigators found that histamine H1 receptor antagonists at relatively low doses facilitate EA analgesia in the acetic acid-induced abdominal writhing test. Investigators aim to further explore whether histamine H1 receptor antagonists also facilitate EA analgesia in humans.The aims of the proposed studies are to: Conduct a clinical trial to demonstrate that H1 receptor antagonists at relatively low doses facilitate EA analgesia in healthy volunteers. This study will recruit 40 healthy normal subjects (aged between 20 and 30 years) who will be randomly assigned to one of four groups: (1) Sham acupuncture (Shallow needling without electrical stimulation) at ST36 and GB34; (2) EA at ST36 and GB34; (3) EA at ST36 and GB34 plus low-dose chlorpheniramine (2 mg); (4) EA at ST36 and GB34 plus regular-dose chlorpheniramine (4 mg). The primary endpoint will be the pain threshold. It is expected that the completion of this proposed study will enhance our knowledge as to how acupuncture analgesia can be promoted by antihistamine drugs given at a low dose and help to define its application for clinical use.

ELIGIBILITY:
Inclusion Criteria:

1. . Age: 20 to 30 years of age.
2. . Agrees to undergo a comprehensive medical history and physical examination.
3. . No history of analgesic, sedative, dietary/appetite medication intake for more than 3 weeks prior to enrolment.

Exclusion Criteria:

1. . An ongoing medical condition that requires active medical intervention or monitoring to avert serious danger to the participant's health or well-being (e.g., hypertension, diabetes mellitus, or epilepsy).
2. . A compromised skin barrier (e.g., skin disease, allergy) that would interfere with the conduct of the EA procedure and assessments of the study.
3. . An implant such as a pacemaker, defibrillator, or electronic medical equipment.
4. . Pregnancy, or planning for pregnancy.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
pain threshold in each group:the current intensity of Transcutaneous electrical stimulation (TCES) | baseline and 10min after treatment
  Transcutaneous electrical stimulation (TCES) is used as a method of inducing pain in the study. The procedure is to attach two electrode patches on the inside of the upper arm of the subject and then connect the electric stimulator. The current intensity will gradually increase from 0 mA, and each time increase 0.5amps until the subject feels pain in the visual analogy. Transcutaneous electrical stimulation (TCES) will be stopped at the visual analog scale of 5 (that means the moderate pain). The current intensity will be compared within and between each group.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hung Chen, PhD, Study Director — Graduate Institute of Acupuncture Science, China Medical University
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Traiffort E, Pollard H, Moreau J, Ruat M, Schwartz JC, Martinez-Mir MI, Palacios JM. Pharmacological characterization and autoradiographic localization of histamine H2 receptors in human brain identified with [125I]iodoaminopotentidine. J Neurochem. 1992 Jul;59(1):290-9. doi: 10.1111/j.1471-4159.1992.tb08903.x. PMID 1351926
- [Background] Zhang WT, Jin Z, Luo F, Zhang L, Zeng YW, Han JS. Evidence from brain imaging with fMRI supporting functional specificity of acupoints in humans. Neurosci Lett. 2004 Jan 2;354(1):50-3. doi: 10.1016/j.neulet.2003.09.080. PMID 14698480
- [Derived] Lee YC, Tu CH, Chung HY, Luo ST, Chu YT, MacDonald IJ, Kotha P, Huang CC, Lane HY, Lin JG, Chen YH. Antihistamine promotes electroacupuncture analgesia in healthy human subjects: A pilot study. J Tradit Complement Med. 2022 Apr 21;12(5):511-517. doi: 10.1016/j.jtcme.2022.04.003. eCollection 2022 Sep. PMID 36081814